CLINICAL TRIAL: NCT05810493
Title: A Cohort of Patients With Phenotyped Diffuse Interstitial Lung Disease With Longitudinal Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Pneumo01
Record Dates: First submitted 2023-03-29; First posted 2023-04-12 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-03

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — Follow-up of disease, therapeutics and evolution

SUMMARY:
The purpose of the study is to conduct a descriptive analysis of the population of patients with an interstitial lung disease received in the pulmonary department of University hospital of Nice (France). Analysis and documentation of clinical forms of the disease, therapeutics used and evolutions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosis of interstitial lung disease according to the multidisciplinary monthly meeting for interstitial lung disease occuring at University hospital of Nice, France

Exclusion Criteria:

* Patient-led opposition to data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ≥ 18 years old; Patients with a formal diagnosis or a provisional diagnosis of interstitial lung disease according to the mutlidisciplinary monthly meeting for interstitial lung disease occuring at University hospital of Nice, France
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Build a retrospective cohort of patients with phenotyped interstitial Lung disease with longitudinal follow-up | 2 years

SECONDARY OUTCOMES:
Follow-up of progression criteria according to diagnosis | 2 years
  Change in pulmonary functional tests
Follow-up of progression criteria according to diagnosis | 2 years
  Change in respiratory symptoms
Follow-up of progression criteria according to diagnosis | 2 years
  Change in High-resolution Computed Tomography (HRCT) images
Follow-up of progression criteria according to diagnosis | 2 years
  Impact of interstitial lung disease treatements

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No